CLINICAL TRIAL: NCT00405834
Title: A Pilot Study of the Envision® Surface in a Patient Population at High Risk for or Who Have Pressure Ulcers: Evaluation of Pressure Ulcer Incidence, Changes in Existing Pressure Ulcers, Clinical Staff Satisfaction and Patient Comfort
Brief Title: A Pilot Study of the Envision® Surface
Status: Completed | Type: Observational
Sponsor: Hill-Rom (Industry)
Responsible Party: Gordon MacFarlane, PhD, Director of Clinical Research, Hill-Rom
Other Study IDs: CR-0065
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2007-06

CONDITIONS: Pressure Ulcers
Keywords: Pressure Ulcers
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Envision® Patient Support System

SUMMARY:
This study is to evaluate the clinical safety and effectiveness of the Envision® surface.

DETAILED DESCRIPTION:
This study is to evaluate the clinical safety and effectiveness of the Envision® surface placed on the TotalCare® frame in pressure ulcer prevention and management, patient comfort, and staff acceptance in the critical care environment

ELIGIBILITY:
Inclusion Criteria:

* Subject weighs between 70 and 400 pounds Subject to remain on Envision Surface for at least 3 days Subject at risk for pressure ulcers (Braden Score < 14) or has existing ulcer of any stage Subject is able to provide voluntary consent

Exclusion Criteria:

* Subject requires pulmonary treatment surface Subject declines consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-06; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Fisher, RN, CWOCN, Study Director — Sinai Hospital of Baltimore / Lifebridge Health
Locations (1):
- Sinai Hospital of Baltimore, Baltimore, Maryland, United States